CLINICAL TRIAL: NCT02513043
Title: Feasibility of Medical Abortion by Direct-to-Consumer Telemedicine
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1031
Record Dates: First submitted 2015-07-24; First posted 2015-07-31 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2020-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: medical abortion — medical abortion

SUMMARY:
This pilot study is designed to obtain preliminary data on the safety, acceptability, and feasibility of direct-to-consumer telemedicine abortion.

DETAILED DESCRIPTION:
The objective of this pilot study is to obtain preliminary data on the safety, acceptability, and feasibility of direct-to-consumer telemedicine abortion.

ELIGIBILITY:
Inclusion Criteria:

* desires abortion

Exclusion Criteria:

* medically ineligible for procedure

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 1470 (Actual)
Dates: Start 2016-03-22; Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 1 year
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Erica Chong, MPH, Principal Investigator — Gynuity Health Projects; Elizabeth Raymond, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (17):
- United States (17):
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Carafem, Washington D.C., District of Columbia
  - Carafem, Atlanta, Georgia
  - The University of Hawaii Women's Options Centers, Honolulu, Hawaii
  - Carafem, Skokie, Illinois
  - Emma Goldman Clinic, Iowa City, Iowa
  - Maine Family Planning, Augusta, Maine
  - Carafem, Chevy Chase, Maryland
  - Planned Parenthood Minnesota, North Dakota, South Dakota, Saint Paul, Minnesota
  - Planned Parenthood of Montana, Billings, Montana
  - Planned Parenthood of the Rocky Mountains, New Mexico, New Mexico
  - Choices Women's Medical Center, Jamaica, New York
  - Maine Family Planning, New York, New York
  - Planned Parenthood Columbia Willamette, Portland, Oregon
  - Oregon Health and Sciences University Women's Health Research Unit, Portland, Oregon
  - Planned Parenthood Columbia Willamette, Washington, Washington
  - Oregon Health and Sciences University Women's Health Research Unit, Washington, Washington